CLINICAL TRIAL: NCT06642896
Title: Quantitative Pupillometry in Brain Injury Children : Variation After Osmotherapy
Acronym: OSMOPUPILLO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0212
Record Dates: First submitted 2024-09-23; First posted 2024-10-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Children Brain Injury
Keywords: brain lesion; pupillometry; assess variation in the percentage of pupillary constriction; children; severe head trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- severe head trauma in children with osmotherapy treatment: Admission to the pediatric intensive care or neurosurgical intensive care unit, pupillometry measurement before and after osmotherapy treatment
  Interventions: Device: pupillometer
- pupillometry measurement in non-cerebral pediatric patients: feasibility of pupillometry in children for different age groups and obtain baseline values for non-neurologically sedated children in 4 age groups from 0 to 17 years of age in intensive care and the operating room
  Interventions: Device: pupillometer

INTERVENTIONS:
Device: pupillometer — describe the feasibility of pupillometry measurements in sedated but non-cerebrosed children in intensive care and the operating room
  Groups: pupillometry measurement in non-cerebral pediatric patients
Device: pupillometer — Pupillometry measurements at 5 and 25 minutes for children treated with osmotherapy, followed by measurements twice a day during hospitalization in the intensive care unit
  Groups: severe head trauma in children with osmotherapy treatment

SUMMARY:
Intracranial hypertension (ICH) is a common and serious complication in children admitted to pediatric intensive care units. It is primarily caused by traumatic brain injury but can also result from brain malformations, brain tumors, or neuro-meningeal infections. Rapid identification of ICH in acute settings is crucial to ensure prompt management and mitigate potential consequences, such as severe neurological sequelae or death.

The assessment of the pupillary light reflex is one of the key clinical parameters used to identify ICH in children with neurological injuries. This clinical sign is correlated with neurological prognosis. During an episode of ICH, regardless of the underlying cause, the oculomotor nerve becomes compressed between the midbrain and the temporal lobe, leading to anisocoria (unequal pupil sizes) and loss of pupillary reactivity. Other factors, such as episodes of ischemia or hypoperfusion in the midbrain, can also contribute to decreased pupillary reactivity.

DETAILED DESCRIPTION:
Traditionally, the pupillary light reflex is assessed using a simple light source, with subjective evaluation by a healthcare professional. However, this method has significant inter- and intra-individual variability. Quantitative pupillometry offers a more objective and reproducible way to evaluate pupillary reactivity. In adults, some parameters are well-known indicators of ICH, such as a constriction velocity of less than 0.6 mm/sec and a constriction percentage below 10%. The constriction percentage can be simplified with the Neurological Pupil index (NPI), which ranges from 0 to 5. An NPI of 4 or 5 is considered to indicate good pupillary reactivity. The two quantitative pupillometers currently on the market (Neurolight, Neuroptics) appear to provide similar data for most variables assessed. However, there are few studies evaluating this tool in pediatric patients with neurological injuries.

One study on quantitative pupillometry found that children with neurological injuries and an intracranial pressure (ICP) above 20 mmHg had significantly lower pupillary reactivity, NPI, constriction percentage, and dilation and constriction velocities compared to children without ICH.

Osmotherapy is a commonly used pharmacological intervention in pediatrics to lower intracranial pressure and improve cerebral perfusion pressure. Based on the work of Freeman et al., we hypothesize that the pupillary constriction percentage improves after osmotherapy in children with neurological injuries.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in a pediatric intensive care unit or neurosurgical intensive care unit
* Inclusion within 24 hours of ICU admission
* with clinically suspected HTIC (disorders of consciousness with transcranial Doppler abnormality, symptoms of involvement, poor cerebral perfusion pressure) for which osmotherapy is prescribed

Exclusion Criteria:

* Presence of eye damage (or antecedent)
* Refusal by parents and/or child Opposition by child or parental guardians.
* Persons not affiliated to the social security system.
* Protected persons (under guardianship, curatorship, pregnant or breast- feeding women, persons deprived of their liberty, persons not subject to a psychiatric measure

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged 1 month to 17 years with brain lesion receiving osmotherapy
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
to describe and evaluate the variation in the percentage of pupillary constriction (CON) before, and after osmotherapy in neuro-injured children. | at 10 days
  Delta (in percentage difference, and in delta of values) of the constriction (CON) between the last available measurement before the osmotherapy was started, and the measurement 5 minutes after the end (at 25 minutes after the start of the osmotherapy).
  For each child, the eye with the lowest constriction (CON) value before osmotherapy will be considered.
Describe the feasibility of pupillometry in children for different age groups, and obtain baseline values for the sedated, non-neurosed child. | at 1 minute and 25 minutes
  Success rate in obtaining pupillometric values for different age groups. Pupillometric values: QPI (quantitative pupillometry index) in intensive care and the operating room
Describe the feasibility of pupillometry in children for different age groups, and obtain baseline values for the sedated, non-neurosed child. | at 1 minute and 25 minutes
  Success rate in obtaining pupillometric values for different age groups. Pupillometric values: latency (LAT) in intensive care and the operating room
Describe the feasibility of pupillometry in children for different age groups, and obtain baseline values for the sedated, non-neurosed child. | at 1 minute and 25 minutes
  Success rate in obtaining pupillometric values for different age groups. Pupillometric values: constriction velocity (ACV) and dilatation velocity (ADV) in mm/sec in intensive care and the operating room
Describe the feasibility of pupillometry in children for different age groups, and obtain baseline values for the sedated, non-neurosed child. | at 1 minute and 25 minutes
  Success rate in obtaining pupillometric values for different age groups. Pupillometric values: minimum (MIN) and maximum (MAX) pupillary diameter in mm in intensive care and the operating room

SECONDARY OUTCOMES:
In the age subgroup of children with an intracranial pressure (ICP) sensor (pathological if ICP more than 20mmHg), evaluate the relationship between intracranial pressure and the various pupillometry values (LAT). | per 12h during 10 days
  Assessing the association between latency in sec (LAT) and ICP (mmhg)
In the age subgroup of children with an intracranial pressure (ICP) sensor (pathological if ICP more than 20mmHg), evaluate the relationship between intracranial pressure and the various pupillometry values (QPI). | per 12h during 10 days
  Assessing the association between measurements of pupillometry, QPI, quantitative pupillometry index
In the age subgroup of children with an intracranial pressure (ICP) sensor (pathological if ICP more than 20mmHg), evaluate the relationship between intracranial pressure and the various pupillometry values.(CON) | per 12h during 10 days
  Assessing the association between measurements of pupillometry, percentage of constriction (CON) and ICP.
In the age subgroup of children with an intracranial pressure (ICP) sensor (pathological if more than 20mmHg), evaluate the relationship between intracranial pressure and the various pupillometry values (Max; Min) | per 12h during 10 days
  To asses association between intracranial pressure and minimum et maximum pupillary diameter (in mm).
In the age subgroup of children with an intracranial pressure (ICP) sensor (pathological if more than 20mmHg), evaluate the relationship between intracranial pressure and the various pupillometry values. (ACV and ADV) | per 12h during 10 days
  To asses association between ICP and pupillometry values : constriction velocity (ACV) and dilatation velocity (ADV) in mm.sec
Comparison of pupillometry values between neuro-sedated and non-neuro-sedated children, adjusting for age | at 1 and 25 minutes
  measurement of pupillometric parameters : latence (in sec)
Comparison of pupillometry values between neuro-sedated and non-neuro-sedated children, adjusting for age. | at 1 and 25 minutes
  measurement of pupillometric parameters : quantitative pupillometry index, pupil constriction
Comparison of pupillometry values between neuro-sedated and non-neuro-sedated children, adjusting for age. | at 1 and 25 minutes
  measurement of pupillometric parameters : Minimum and maximum pupillary diameter (in mm)
Comparison of pupillometry values between neuro-sedated and non-neuro-sedated children, adjusting for age. | at 1 and 25 min
  measurement of pupillometric parameters constriction velocity (ACV), dilatation velocity (ADV) in mm/sec
Describe the evolution of different pupillometry measurements before and after osmotherapy | at 15 , 25, 35, 45, 60, 120, 240 minutes
  Measure of pupillometry: CON and QPI after osmotherapy administration
Describe the evolution of different pupillometry measurements before and after osmotherapy | [Time Frame: at 15 , 25, 35, 45, 60, 120, 240 minutes]
  Measure of pupillometry : constriction velocity (ACV), dilatation velocity (ADV) in mm/sec
Describe the evolution of different pupillometry measurements before and after osmotherapy | [Time Frame: at 15 , 25, 35, 45, 60, 120, 240 minutes]
  Measure of pupillometry: latence (in mm)
Describe the evolution of different pupillometry measurements before and after osmotherapy | at 15 , 25, 35, 45, 60, 120, 240 minutes
  Measure of pupillometry: Min and max pupillary diameter in mm.
Assessing the relationship between transcranial Doppler (CTD) results: pulsatility index (PI) and diastolic velocity (Vd) | 2 times a day for 10 days or on discharge from hospital
  Repeated pupillometry measurements : (LAT) latence in sec and transcranial doppler
Assessing the relationship between transcranial Doppler (CTD) results: pulsatility index (PI) and diastolic velocity (Vd) | 2 times a day for 10 days or on discharge from hospital
  Repeated pupillometry measurements QPI and CON and transcranial doppler
Assessing the relationship between transcranial Doppler (CTD) results: pulsatility index (PI) and diastolic velocity (Vd) | 2 times a day for 10 days or on discharge from hospital
  Repeated pupillometry measurements (Maximum and minimum pupillary diameter in mm) and transcranial doppler
Assessing the relationship between transcranial Doppler (CTD) results: pulsatility index (PI) and diastolic velocity (Vd) | 2 times a day for 10 days or on discharge from hospital
  Repeated pupillometry measurements (constriction velocity (ACV) and dilatation velocity (ADV) in mm.sec) and transcranial doppler

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Grenoble Alpes, Grenoble, ISERE
  - Grenoble Alpes University Hospital, La Tronche

IPD SHARING:
Plan to Share IPD: No
This is an observational study, which does not modify the management of children with brain lesions, nor does it generate additional therapies.

REFERENCES:
- [Background] Winston M, Zhou A, Rand CM, Dunne EC, Warner JJ, Volpe LJ, Pigneri BA, Simon D, Bielawiec T, Gordon SC, Vitez SF, Charnay A, Joza S, Kelly K, Panicker C, Rizvydeen S, Niewijk G, Coleman C, Scher BJ, Reed DW, Hockney SM, Buniao G, Stewart T, Trojanowski L, Brogadir C, Price M, Kenny AS, Bradley A, Volpe NJ, Weese-Mayer DE. Pupillometry measures of autonomic nervous system regulation with advancing age in a healthy pediatric cohort. Clin Auton Res. 2020 Feb;30(1):43-51. doi: 10.1007/s10286-019-00639-3. Epub 2019 Sep 25. PMID 31555934
- [Background] Boev AN, Fountas KN, Karampelas I, Boev C, Machinis TG, Feltes C, Okosun I, Dimopoulos V, Troup C. Quantitative pupillometry: normative data in healthy pediatric volunteers. J Neurosurg. 2005 Dec;103(6 Suppl):496-500. doi: 10.3171/ped.2005.103.6.0496. PMID 16383247
- [Background] Rouche O, Wolak-Thierry A, Destoop Q, Milloncourt L, Floch T, Raclot P, Jolly D, Cousson J. Evaluation of the depth of sedation in an intensive care unit based on the photo motor reflex variations measured by video pupillometry. Ann Intensive Care. 2013 Feb 22;3(1):5. doi: 10.1186/2110-5820-3-5. PMID 23433043
- [Background] Freeman AD, McCracken CE, Stockwell JA. Automated Pupillary Measurements Inversely Correlate With Increased Intracranial Pressure in Pediatric Patients With Acute Brain Injury or Encephalopathy. Pediatr Crit Care Med. 2020 Aug;21(8):753-759. doi: 10.1097/PCC.0000000000002327. PMID 32195898
- [Background] Robba C, Moro Salihovic B, Pozzebon S, Creteur J, Oddo M, Vincent JL, Taccone FS. Comparison of 2 Automated Pupillometry Devices in Critically III Patients. J Neurosurg Anesthesiol. 2020 Oct;32(4):323-329. doi: 10.1097/ANA.0000000000000604. PMID 31033624
- [Background] Bower MM, Sweidan AJ, Xu JC, Stern-Neze S, Yu W, Groysman LI. Quantitative Pupillometry in the Intensive Care Unit. J Intensive Care Med. 2021 Apr;36(4):383-391. doi: 10.1177/0885066619881124. Epub 2019 Oct 10. PMID 31601157
- [Background] Ritter AM, Muizelaar JP, Barnes T, Choi S, Fatouros P, Ward J, Bullock MR. Brain stem blood flow, pupillary response, and outcome in patients with severe head injuries. Neurosurgery. 1999 May;44(5):941-8. doi: 10.1097/00006123-199905000-00005. PMID 10232526
- [Background] Manley GT, Larson MD. Infrared pupillometry during uncal herniation. J Neurosurg Anesthesiol. 2002 Jul;14(3):223-8. doi: 10.1097/00008506-200207000-00009. PMID 12172296
- [Background] Rameshkumar R, Bansal A, Singhi S, Singhi P, Jayashree M. Randomized Clinical Trial of 20% Mannitol Versus 3% Hypertonic Saline in Children With Raised Intracranial Pressure Due to Acute CNS Infections. Pediatr Crit Care Med. 2020 Dec;21(12):1071-1080. doi: 10.1097/PCC.0000000000002557. PMID 33003179
- [Background] Piper BJ, Harrigan PW. Hypertonic saline in paediatric traumatic brain injury: a review of nine years' experience with 23.4% hypertonic saline as standard hyperosmolar therapy. Anaesth Intensive Care. 2015 Mar;43(2):204-10. doi: 10.1177/0310057X1504300210. PMID 25735686
- [Background] Kochanek PM, Adelson PD, Rosario BL, Hutchison J, Miller Ferguson N, Ferrazzano P, O'Brien N, Beca J, Sarnaik A, LaRovere K, Bennett TD, Deep A, Gupta D, Willyerd FA, Gao S, Wisniewski SR, Bell MJ; ADAPT Investigators. Comparison of Intracranial Pressure Measurements Before and After Hypertonic Saline or Mannitol Treatment in Children With Severe Traumatic Brain Injury. JAMA Netw Open. 2022 Mar 1;5(3):e220891. doi: 10.1001/jamanetworkopen.2022.0891. PMID 35267036
- [Background] Rallis D, Poulos P, Kazantzi M, Chalkias A, Kalampalikis P. Effectiveness of 7.5% hypertonic saline in children with severe traumatic brain injury. J Crit Care. 2017 Apr;38:52-56. doi: 10.1016/j.jcrc.2016.10.014. Epub 2016 Oct 21. PMID 27838440
- [Background] Melo JR, Di Rocco F, Blanot S, Cuttaree H, Sainte-Rose C, Oliveira-Filho J, Zerah M, Meyer PG. Transcranial Doppler can predict intracranial hypertension in children with severe traumatic brain injuries. Childs Nerv Syst. 2011 Jun;27(6):979-84. doi: 10.1007/s00381-010-1367-8. Epub 2011 Jan 5. PMID 21207041
- See also: Epidemiology of head injuries in France and other Western countries — https://www.santepubliquefrance.fr/docs/epidemiologie-des-traumatismes-craniens-en-france-et-dans-les-pays-occidentaux-synthese-bibliographique-avril-2016
- See also: intracranial hypertension in infants — https://www.pediatrie-pratique.com/journal/article/l-hypertension-intracranienne-du-nourrisson-0